CLINICAL TRIAL: NCT07002463
Title: "Comparison of Outcomes of Physiotherapist- and Robot-Assisted Upper Limb Therapy and Their Association With Muscle Tone and Motor Function in Subacute Stroke Patients"
Brief Title: "Comparison of Therapist-Led and Robot-Assisted Arm Therapy in Subacute Stroke Rehabilitation"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Responsible Party: Principal Investigator, Denis Moskiewicz, M.Sc., Assistant Lecturer, Dept. of Neurological and Pediatric Physiotherapy, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LUNA-AWF-2025-01
Record Dates: First submitted 2025-05-22; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Hemiparesis; Muscle Spasticity; Upper Extremity Dysfunction; Subacute Stroke
MeSH Terms: conditions — Stroke; Paresis; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two parallel groups: (1) robot-assisted upper limb rehabilitation using Luna EMG or (2) therapist-assisted upper limb rehabilitation. Both groups also receive the same standard rehabilitation program. Randomization was performed using simple urn-based drawing by an individual independent of the study team. An additional balancing step was applied post-assignment to ensure equal group sizes. Interventions are delivered in parallel over 6 weeks, 5 days per week.
Who Masked: Outcomes Assessor
Masking Description: Only the outcomes assessor is blinded. Functional and quality of life assessments (e.g., FMA-UE, Box and Blocks Test, EQ-5D-5L) are conducted by an independent physiotherapist who is not involved in treatment delivery and remains unaware of the participants' group assignments.
  Due to the nature of the intervention, participants are aware of their treatment allocation (robot-assisted vs. therapist-assisted training). Similarly, physiotherapists delivering the robotic or therapist-assisted upper limb training (based on 50 EMG-triggered or assisted repetitions) are necessarily aware of group allocation. However, physiotherapists delivering the standard rehabilitation program (common to both groups) are not informed about group assignment and are considered blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-assisted training (Luna EMG) (Experimental): A robotic rehabilitation device using EMG-triggered movement assistance for upper limb recovery after stroke.
  Interventions: Device: Luna EMG
- Therapist-assisted training (Active Comparator): A physiotherapist assists the participant in performing 4 specific upper limb movements (50 repetitions each), matching the robotic training protocol.
  Interventions: Behavioral: Therapist-assisted upper limb training

INTERVENTIONS:
Device: Luna EMG — Participants receive additional upper limb rehabilitation using the Luna EMG robotic system. Each session includes 4 EMG-triggered exercises (shoulder flexion, external rotation, elbow extension, and forearm supination), with 50 repetitions per movement. The intervention is delivered 5 days per week for 6 weeks alongside a standard rehabilitation program.
  Arms: Robot-assisted training (Luna EMG)
Behavioral: Therapist-assisted upper limb training — Participants receive additional upper limb rehabilitation with a physiotherapist performing assisted movements equivalent to the robotic training protocol. Each session includes 4 assisted exercises (shoulder flexion, external rotation, elbow extension, and forearm supination), with 50 repetitions per movement. The intervention is delivered 5 days per week for 6 weeks alongside a standard rehabilitation program.
  Arms: Therapist-assisted training

SUMMARY:
This study aims to compare the outcomes of upper limb motor therapy conducted by a physiotherapist with robot-assisted therapy using the Luna EMG device in patients in the subacute phase after stroke. Additionally, the study will examine the correlation between changes in muscle tone and motor function improvement. The randomized controlled trial will be conducted at the Rehabilitation Department of the T. Marciniak Lower Silesian Specialist Hospital in Wrocław, Poland. Two groups (robot-assisted vs. conventional therapy) will perform identical sets of movements with matched repetition counts over a 6-week therapy period. Functional improvement will be assessed using Fugl-Meyer Upper Extremity Assessment (FMA-UE), Box and Block Test (B&BT), EQ-5D-5L, and MyotonPro measurements.

DETAILED DESCRIPTION:
Stroke often leads to upper limb motor impairment, spasticity, and reduced independence. Robot-assisted rehabilitation, including devices like Luna EMG, may increase therapy intensity and patient motivation through feedback and movement intention detection via EMG signals.

This interventional study includes 50 participants post-stroke, randomly assigned to either robot-assisted therapy (Luna EMG) or conventional physiotherapist-led therapy. Both groups receive standard rehabilitation (75 minutes/day), with an additional 45-minute targeted upper limb training session. Sessions are conducted 5 days a week for 6 weeks.

Muscle tone will be assessed using the Modified Ashworth Scale and biomechanical parameters (stiffness, oscillation) with MyotonPro. Motor performance will be evaluated using the Fugl-Meyer Assessment (FMA-UE) and the Box and Block Test (B&BT). Quality of life and pain perception will also be measured using the EQ-5D-5L and a numeric rating scale (NRS).

Outcome measures will be collected at baseline, after 3 weeks, after 6 weeks of therapy, and 3 weeks post-intervention to evaluate both immediate and short-term effects of the intervention. This study seeks to identify whether robotic rehabilitation offers measurable advantages over traditional methods in early post-stroke recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90
* First-ever ischemic or hemorrhagic stroke within 6 weeks prior to enrollment
* Stable medical condition
* Fugl-Meyer Assessment for Upper Extremity (FMA-UE) ≤ 94
* Mini-Mental State Examination (MMSE) ≥ 23
* Signed informed consent

Exclusion Criteria:

* Fixed contractures in upper limb
* MAS ≥ 3 in any upper limb muscle
* Severe vision/hearing problems
* Severe dysphagia or respiratory issues
* Myasthenia or myasthenic syndrome

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment for Upper Extremity (FMA-UE) | Baseline, Week 3, Week 6, and 3 weeks after therapy completion
  Functional motor recovery of the affected upper limb, scored 0-66 (or 94, depending on version used). Higher scores indicate better function.

SECONDARY OUTCOMES:
Box and Blocks Test (B&BT) | Baseline, Week 3, Week 6, and 3 weeks after therapy completion
  Measures gross manual dexterity by counting the number of blocks transferred in 60 seconds.
  Higher scores indicate better manual dexterity.
EQ-5D-5L | Baseline, Week 3, Week 6, and 3 weeks after therapy completion
  Quality of life across 5 domains (mobility, self-care, usual activities, pain/discomfort, anxiety/depression).
  Scores are reported on a scale from 0 to 1, where 0 represents the worst possible health state and 1 represents the best possible health state. Higher scores indicate better quality of life.
Muscle Tone - Modified Ashworth Scale (MAS) | Baseline, Week 3, Week 6, and 3 weeks after therapy completion
  Spasticity of upper limb muscles scored 0-4. It scores resistance during passive soft-tissue stretching on a scale from 0 to 4.
  The scale is as follows:
  0 = No increase in muscle tone
  1 = Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion
  1+ = Slight increase in muscle tone, manifested by a catch followed by minimal resistance throughout the remainder (less than half) of the range of motion 2 = More marked increase in muscle tone through most of the range of motion, but affected part(s) easily moved 3 = Considerable increase in muscle tone, passive movement difficult 4 = Affected part(s) rigid in flexion or extension Higher scores indicate greater spasticity (worse outcome).
Muscle Oscillation Frequency Measured by MyotonPRO | Baseline, Week 3, Week 6, and 3 weeks after therapy completion
  Objective measurement of natural oscillation frequency (Hz) of selected upper limb muscles using the MyotonPRO device. This parameter reflects muscle tone and viscoelastic properties. Higher values indicate increased muscle tone.
Muscle Stiffness Measured by MyotonPRO | Baseline, Week 3, Week 6, and 3 weeks after therapy completion
  Objective measurement of muscle stiffness (N/m) in selected upper limb muscles using the MyotonPRO device. Stiffness represents resistance to deformation. Higher values indicate greater muscle rigidity.
Muscle Elasticity Measured by MyotonPRO | Baseline, Week 3, Week 6, and 3 weeks after therapy completion
  Measurement of muscle elasticity (logarithmic decrement) in selected upper limb muscles using the MyotonPRO device. Lower values indicate more elastic (less stiff) muscle tissue.
Muscle Relaxation Time Measured by MyotonPRO | Baseline, Week 3, Week 6, and 3 weeks after therapy completion
  Measurement of muscle relaxation time (milliseconds) in selected upper limb muscles using the MyotonPRO device. This is the time taken for the muscle to return to its initial state after deformation. Shorter relaxation time suggests better muscle function.
Muscle Creep Measured by MyotonPRO | Baseline, Week 3, Week 6, and 3 weeks after therapy completion
  Assessment of muscle creep (deformation over time under constant load) in selected upper limb muscles using the MyotonPRO device. Higher creep values indicate greater viscoelastic deformation.
Pain Intensity (NRS 0-10) | Baseline, Week 3, Week 6, and 3 weeks after therapy completion (Rest and activity)
  Numeric pain rating scale (0 = no pain, 10 = worst imaginable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Denis Moskiewicz, M.Sc., Study Chair — Department of Physiotherapy, Wroclaw University of Health and Sport Sciences, 51-612 Wrocław, Poland
Locations (1):
- Lower Silesian Specialist Hospital T. Marciniak - Emergency Medicine Center, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Yes